CLINICAL TRIAL: NCT05877469
Title: Effects of Mat Pilates Versus Functional Training on Pain, Range of Motion and Disability in Mechanical Low Back Pain
Brief Title: Effects of MAT Pilates Versus Functional Training on Mechanical Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC//23/0107/Wasifa Haider
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Mechanical Low Back Pain
Keywords: Disability; pilates Training; Range of motion; Pain
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mat pilates training group (Active Comparator): Mat pilates training involve leg lifts, toe taps, Single leg stretch, one leg circle, side bend preparation, side kicks, side leg lifts, swan dive, hovers, roll down, crisscross and planks. Treatments will be provided in 30 mins, three sessions per week for 8 consecutive weeks.
  Interventions: Other: Mat pilates Training
- Functional training group (Experimental): Functional training involve glute bridge, squats, pushups, lateral lunge, step up to shoulder press, goblet squats and woodchop. Treatments will be provided in 30 mins, three sessions per week for 8 consecutive weeks.
  Interventions: Other: Functional Training

INTERVENTIONS:
Other: Mat pilates Training — In this group 22 patients will perform mat pilates training. Patients will be asked to stay comfortable while performing mat pilates exercies that involve different types of movements of whole body like leg lifts, toe taps, Single leg stretch, one leg circle, side bend preparation, side kicks, side leg lifts, roll down and crisscross to improve the core strength. Treatments will be provided in 30 mins, three sessions per week for 8 consecutive weeks.
  Arms: mat pilates training group
Other: Functional Training — In this group 22 patients will perform functional training. Patients will be instructed to perform their daily living movements like squatting, reaching, or even carrying a heavy object. These exercises typically use the whole body and emphasize core strength and stability. Functional training typically uses weight-bearing activities that work the core muscles in the torso. the functional movements include involve glute bridge, squats, pushups, lateral lunge, step up to shoulder press, goblet and squats. Treatments will be provided in 30 mins, three sessions per week for 8 consecutive weeks.
  Arms: Functional training group

SUMMARY:
This study will be a randomized clinical trial. Total 44 Subjects with mechanical low back pain will be assigned randomly by using non probability convenient random sampling in to two groups with 22 subjects in each group. Subjects in one group will be treated with mat Pilates training and the other group with the functional training. NPRS, Inclinometer and urdu version of Modified Oswestry Disablility questionair would be used to measure the outcome of pain, Range of Motion and Disability respectively. After data collection from defined study setting, data will be entered and analyzed at Riphah International University lahore.

DETAILED DESCRIPTION:
Mechanical low back pain refers to back pain that arises intrinsically from the spine, intervertebral disks, or surrounding soft tissues. This includes lumbosacral muscle strain, disk herniation, lumbar spondylosis, spondylolisthesis, spondylolysis, vertebral compression fractures, and acute or chronic traumatic injury. Repetitive trauma and overuse are common causes of chronic mechanical low back pain, which is often secondary to workplace injury. Pilates focus is improving the core strength, it trains the body as an integrated whole. Functional training involves the daily life activities that also targets on core stability and strength.

The aim of the study is to present the current state of knowledge concerning the application of pilates and functional training in terms of duration, frequency and specific exercises in the management of mechanical low back pain in terms of pain, ROM and disability improvement.

Effects of Mat Pilates and functional training on mechanical low back pain are checked individually before but their effects are not compared previously.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Age group 25-40
* Patient having mechanical low back pain for more than 12 weeks

Exclusion Criteria:

* Pregnancy
* Previous spinal surgery
* Orthopedic and neurological diseases
* Patients with serious spinal pathologies( tumor, fracture and autoimmune conditions)

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Modified Oswestry LBP disability index | 3 weeks
  MODI consists of 10 items questioning daily life activities. These are; pain severity, personal care, lifting, walking, sitting, standing, sleeping, social life, travel and pain. There are 6 options between 0-5 points for each item. Zero indicates mild case, 5 indicates worst case, 0-14 weak, 15-29 moderate, 30 above the functional limit
Numeric Pain Rating Scale | 3 weeks
  NPRS consists of a scale with 0-10 readings. The zero denotes no pain while 1, 2, 3 denotes to mild pain, 4, 5, 6 denotes to moderate pain while 7-10 denotes to severe pain.
Inclinometer | 3 weeks
  Inclinometer is used to measure range of motion of lumber flexion, extension and left/Right side bending

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad sanaullah, MS, Principal Investigator — Riphah International University
Locations (1):
- District Headquarter Hospital Sahiwal, Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Will JS, Bury DC, Miller JA. Mechanical Low Back Pain. Am Fam Physician. 2018 Oct 1;98(7):421-428. PMID 30252425
- [Background] Stevans JM, Delitto A, Khoja SS, Patterson CG, Smith CN, Schneider MJ, Freburger JK, Greco CM, Freel JA, Sowa GA, Wasan AD, Brennan GP, Hunter SJ, Minick KI, Wegener ST, Ephraim PL, Friedman M, Beneciuk JM, George SZ, Saper RB. Risk Factors Associated With Transition From Acute to Chronic Low Back Pain in US Patients Seeking Primary Care. JAMA Netw Open. 2021 Feb 1;4(2):e2037371. doi: 10.1001/jamanetworkopen.2020.37371. PMID 33591367
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Background] Urits I, Burshtein A, Sharma M, Testa L, Gold PA, Orhurhu V, Viswanath O, Jones MR, Sidransky MA, Spektor B, Kaye AD. Low Back Pain, a Comprehensive Review: Pathophysiology, Diagnosis, and Treatment. Curr Pain Headache Rep. 2019 Mar 11;23(3):23. doi: 10.1007/s11916-019-0757-1. PMID 30854609
- [Background] Yalfani A, Raeisi Z, Koumasian Z. Effects of eight-week water versus mat pilates on female patients with chronic nonspecific low back pain: Double-blind randomized clinical trial. J Bodyw Mov Ther. 2020 Oct;24(4):70-75. doi: 10.1016/j.jbmt.2020.06.002. Epub 2020 Jun 27. PMID 33218568
- [Background] Paolucci T, Attanasi C, Cecchini W, Marazzi A, Capobianco SV, Santilli V. Chronic low back pain and postural rehabilitation exercise: a literature review. J Pain Res. 2018 Dec 20;12:95-107. doi: 10.2147/JPR.S171729. eCollection 2019. PMID 30588084
- [Background] Cortell-Tormo JM, Sanchez PT, Chulvi-Medrano I, Tortosa-Martinez J, Manchado-Lopez C, Llana-Belloch S, Perez-Soriano P. Effects of functional resistance training on fitness and quality of life in females with chronic nonspecific low-back pain. J Back Musculoskelet Rehabil. 2018 Feb 6;31(1):95-105. doi: 10.3233/BMR-169684. PMID 28826168
- [Background] Batibay S, Kulcu DG, Kaleoglu O, Mesci N. Effect of Pilates mat exercise and home exercise programs on pain, functional level, and core muscle thickness in women with chronic low back pain. J Orthop Sci. 2021 Nov;26(6):979-985. doi: 10.1016/j.jos.2020.10.026. Epub 2020 Dec 29. PMID 33386201
- [Background] O'Keeffe M, O'Sullivan P, Purtill H, Bargary N, O'Sullivan K. Cognitive functional therapy compared with a group-based exercise and education intervention for chronic low back pain: a multicentre randomised controlled trial (RCT). Br J Sports Med. 2020 Jul;54(13):782-789. doi: 10.1136/bjsports-2019-100780. Epub 2019 Oct 19. PMID 31630089
- [Background] Eliks M, Zgorzalewicz-Stachowiak M, Zenczak-Praga K. Application of Pilates-based exercises in the treatment of chronic non-specific low back pain: state of the art. Postgrad Med J. 2019 Jan;95(1119):41-45. doi: 10.1136/postgradmedj-2018-135920. Epub 2019 Jan 12. PMID 30636192
- [Background] Tsauo JY, Chen WH, Liang HW, Jang Y. The effectiveness of a functional training programme for patients with chronic low back pain--a pilot study. Disabil Rehabil. 2009;31(13):1100-6. doi: 10.1080/09638280802511047. PMID 19802926
- [Background] Amaral DDV, Miyamoto GC, Franco KFM, Dos Santos Franco YR, Bastos De Oliveira NT, Hancock MJ, Van Tulder MW, Nunes Cabral CM. Examination of a Subgroup of Patients With Chronic Low Back Pain Likely to Benefit More From Pilates-Based Exercises Compared to an Educational Booklet. J Orthop Sports Phys Ther. 2020 Apr;50(4):189-197. doi: 10.2519/jospt.2019.8839. Epub 2019 Aug 23. PMID 31443627
- [Background] Amjad F, Mohseni-Bandpei MA, Gilani SA, Ahmad A, Waqas M, Hanif A. Urdu version of Oswestry disability index; a reliability and validity study. BMC Musculoskelet Disord. 2021 Mar 29;22(1):311. doi: 10.1186/s12891-021-04173-0. PMID 33781267
- [Background] Neeley DK, George SZ, Minick K, Snow G, Brennan G. Four Variables Were Sufficient for Low Back Pain: Determining Which Patient-Reported Tools Pain and Disability Improvements. J Orthop Sports Phys Ther. 2022 Oct;52(10):685-693. doi: 10.2519/jospt.2022.11018. Epub 2022 Aug 12. PMID 35960508
- [Background] Sedrez JA, Furlanetto TS, Gelain GM, Candotti CT. Validity and Reliability of Smartphones in Assessing Spinal Kinematics: A Systematic Review and Meta-analysis. J Manipulative Physiol Ther. 2020 Jul-Aug;43(6):635-645. doi: 10.1016/j.jmpt.2019.10.012. Epub 2020 Sep 6. PMID 32900546